CLINICAL TRIAL: NCT05746104
Title: Intraoperative Molecular Imaging of Central Nervous System Tumors Using Same Day Second Window Imaging With Indocyanine Green (TumorGlow™ - CNS)
Brief Title: Second Window Indocyanine Green for All Nervous System Tumors
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UPCC 14321; 850516 (Other: University of Pennsylvania)
Record Dates: First submitted 2023-02-17; First posted 2023-02-27 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Nervous System Tumor
MeSH Terms: conditions — Nervous System Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- SWIG Arm (Experimental): This is the only arm for the study and will be experimental. All patients will receive the appropriate dosage of the study drug, which will then be used for visualization of the tumor intraoperatively.
  Interventions: Drug: Administration of Indocyanine Green (ICG) and Visualization of Tumor

INTERVENTIONS:
Drug: Administration of Indocyanine Green (ICG) and Visualization of Tumor — A single dose of the study drug, ICG, of less than 2 mg/kg will be administered on the day of surgery. The visualization of second window ICG for tumor will be performed approximately one to four hours after administration, depending on how long it takes for the neurosurgeon to get through the skin/skull or lamina/dura to the tumor.

SUMMARY:
The study is being conducted to determine if a same-day, low-dose intravenous (into a vein) injection of indocyanine green (ICG) (FDA-approved dye) being detected by using an imaging system can be a useful tool in identifying and differentiating tumor tissue from normal tissues.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients 18 years of age and older
2. Patients presenting with a nervous system tumor presumed to be resectable and at risk for local recurrence on pre-operative assessment
3. Good operative candidates, as determined by the treating physician and multidisciplinary team
4. Subjects capable of giving informed consent

Exclusion Criteria:

1. Pregnant women, as determined by urinary or serum beta hCG within 48 hours of surgery
2. Subjects with a history of iodide allergies
3. Vulnerable patient populations
4. Patients unable to participate in the consent process
5. Patients with history of uncontrolled HTN (requiring ER admission or ≥ 3 BP medications)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2027-02-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Tumor NIR Signal Compared to Background Brain Normal Signal (SBR) | Surgery
  SBR analysis will be stratified by histology, and the dosing and timing flowchart will be used to achieve optimal SBR.
NIR Efficiency | Surgery
  After examining the "equivocal tissue" with white light and NIR imaging, a per person success will be recorded, if least one additional specimen is resected using NIR. NIR will be considered efficacious, if significantly more than 10% of patients meet the success criteria. Each histology will be tested separately.
NIR True Positive Rate | Surgery
  Of the additionally resected specimens using NIR, we will find the true positive rate based on pathology. The entire sample will be evaluated jointly; then, each histology will be evaluated separately as there may be multiple specimens per patient surgery. NIR will be considered efficacious if the true positive rate is significantly greater than 50%.

SECONDARY OUTCOMES:
Safety and Toxicity | Surgery
  Safety and toxicity will be evaluated by review of vital signs and any reported or observed adverse events (AEs).
Association Between Resection Decision and Pathology | Surgery
  Test for an association between a change in resection decision (yes/no) and the pathology results for all resected equivocal tissues will be completed. The association will be tested unadjusted and after controlling tumor location stratified by histology.
Sensitivity | Surgery
  The ROC curve will be analyzed, and the sensitivity, with its respective confidence intervals, will be estimated.
Specificity | Surgery
  The ROC curve will be analyzed, and the specificity, with their respective confidence intervals, will be estimated.
Positive Predictive Value | Surgery
  The ROC curve will be analyzed, and the positive predictive value, with their respective confidence intervals, will be estimated.
Negative Predictive Value | Surgery
  The ROC curve will be analyzed, and the negative predictive value, with their respective confidence intervals, will be estimated.

CONTACTS AND LOCATIONS:
Locations (1):
- Pennsylvania Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No